CLINICAL TRIAL: NCT01662934
Title: A Randomized, Sham Device Controlled, Single Blinded Trial of Portable Transcutaneous Electrical Nerve Stimulation and Heat Therapy Machine in Women With Dysmenorrhea
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUBH_GO_004
Record Dates: First submitted 2012-08-07; First posted 2012-08-13 (Estimated); Last update posted 2013-03-15 (Estimated); Status verified 2013-03

CONDITIONS: Dysmenorrhea
Keywords: dysmenorrhea; transcutaneous electrical nerve stimulation; heat therapy
MeSH Terms: conditions — Dysmenorrhea; Hyperthermia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Sham Comparator): Using not functioning device
  Interventions: Device: sham
- Experimental (Experimental): Using functioning device
  Interventions: Device: I RUNE

INTERVENTIONS:
Device: I RUNE
  Other Names: Transcutaneous electrical nerve stimulation and heat therapy machine
  Arms: Experimental
Device: sham
  Other Names: sham device
  Arms: Sham

SUMMARY:
The hypothesis is that a transcutaneous electrical nerve stimulation and heat therapy machine could reduce dysmenorrhea in women with primary or secondary dysmenorrhea.

DETAILED DESCRIPTION:
Inclusion/Exclusion: Described in Eligibility section. Outcome measures: Change of VAS score before and after use of TENS and heat therapy machine.

ELIGIBILITY:
Inclusion

* Age>19
* Premenopausal
* Moderate or severe dysmenorrhea, mainly in low abdomen area

Exclusion

* Pregnant
* Surgery history on lower abdomen
* Recent history of cancer
* TENS device use is contraindicated
* Ibuprofen use is contraindicated

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Change of VAS before and after application of machine | Immediately before application of machine and 20minutes after application of machine
  Measure the change% of VAS between before application of machine (T0) and 20 minutes after application of machine (T20) in every episode of dysmenorrhea during 1 menstrual cycle The mean of change% of VAS is primary outcome measure

SECONDARY OUTCOMES:
BPI score | 2nd day of menstrual cycle
  Brief Pain Inventory score

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyenggi Do, South Korea

REFERENCES:
- [Derived] Lee B, Hong SH, Kim K, Kang WC, No JH, Lee JR, Jee BC, Yang EJ, Cha EJ, Kim YB. Efficacy of the device combining high-frequency transcutaneous electrical nerve stimulation and thermotherapy for relieving primary dysmenorrhea: a randomized, single-blind, placebo-controlled trial. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:58-63. doi: 10.1016/j.ejogrb.2015.08.020. Epub 2015 Aug 22. PMID 26340453